CLINICAL TRIAL: NCT07201259
Title: Exploring Gut Microbiome Differences in Female Cancer Patients With Varied Ovarian Function and Fertility Outcomes Following Immune Checkpoint Inhibitor Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Shengtao Zhou, Professor, Chief Physician, West China Second University Hospital
Other Study IDs: 2025（1695）
Record Dates: First submitted 2025-08-28; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Malignant Tumors
Keywords: immune checkpoint inhibitors, female, ovarian function, fertility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, feces. Blood samples will be used to monitor serum hormone levels, and stool samples will be used for metagenomic sequencing. These samples will be destroyed after use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICI or ICI combined treatment: Inclusion criteria:
  1. Informed consent must be obtained and documented at the research center prior to initiating any trial procedures.
  2. Female patients aged 18-38 years.
  3. Patients with histologically confirmed solid tumors or soft tissue sarcomas diagnosed via open surgery, laparoscopic surgery, or core needle biopsy.
  4. Patients scheduled to receive ICIs therapy or combination therapy including ICIs;
  5. Normal ovarian function and fertility prior to treatment, defined as regular menstrual cycles, normal serum FSH, LH, E2, P, and AMH levels, and normal gynecological ultrasound findings;
  6. No use of sex hormone medications within 6 months prior to enrollment, including but not limited to estrogens, anti-estrogens hormones, hormonal contraceptives, etc.;
  7. No use of antibiotics or probiotics within 3 months prior to enrollment;
  8. Availability of blood and stool specimens before and after
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
The goal of this observational study is to evaluate the impact of Immune Checkpoint Inhibitor (ICI) treatment on ovarian function and fertility, and to explore the role of gut microbiota in female cancer patients of reproductive age (18-38 years) receiving ICI therapy. The main questions it aims to answer are:

Does ICI treatment alter serum hormone levels (FSH, LH, E2, P, AMH) associated with ovarian function and fertility?

Are there differences in gut microbiota composition and metabolites between patients with different ovarian function and fertility outcomes after ICI treatment?

What are the potential mechanisms by which gut microbiota influences ovarian function and fertility in patients receiving ICIs?

Researchers will compare patients with preserved ovarian function versus those with impaired ovarian function after ICI treatment to identify differences in gut microbiota and metabolic profiles.

Participants will:

Provide blood samples (10 ml per collection) at enrollment and after each of the 6 treatment cycles for hormone level testing and potential future analyses.

Provide stool samples at the same time points for gut microbiota metagenomic sequencing and metabolite analysis.

Undergo regular clinical assessments and follow-ups as part of their standard ICI treatment.

ELIGIBILITY:
Inclusion Criteria:

Collect serum hormone levels post-ICIs treatment to observe the impact of ICIs therapy on female patients.

* Informed consent must be obtained and documented at the research center prior to initiating any trial procedures.
* Female patients aged 18-38 years.
* Patients with histologically confirmed solid tumors or soft tissue sarcomas diagnosed via open surgery, laparoscopic surgery, or core needle biopsy.
* Patients scheduled to receive ICIs therapy or combination therapy including ICIs;
* Normal ovarian function and fertility prior to treatment, defined as regular menstrual cycles, normal serum FSH, LH, E2, P, and AMH levels, and normal gynecological ultrasound findings;
* No use of sex hormone medications within 6 months prior to enrollment, including but not limited to estrogens, anti-estrogens hormones, hormonal contraceptives, etc.;
* No use of antibiotics or probiotics within 3 months prior to enrollment;
* Availability of blood and stool specimens before and after treatment, with the subject's consent to provide these specimens to the central laboratory for study purposes, including but not limited to: i. Potential gut microbiota-related research. ii. Potential metabolite-related research;
* Expected survival >12 weeks;
* ECOG performance status 0-2;
* Adequate organ function, including:
* Bone marrow function: Neutrophil count ≥1500/µL; Platelet count ≥100,000/ µL; Hemoglobin ≥10g/dL
* Liver function: Total bilirubin ≤1.5 times upper limit of normal (ULN) or direct bilirubin ≤1.0 times ULN; AST and ALT ≤2.5 times ULN, must be ≤5 times ULN if liver metastases present
* Renal function: Serum creatinine ≤1.5 times ULN, or creatinine clearance

  * 60 mL/min (calculated using Cockcroft-Gault formula) ;
* Understand the trial protocol and have the ability to comply with the trial plan throughout its duration, including cooperating with any required treatments, examinations, tests, follow-ups, and questionnaires;
* Patient is willing to cooperate with ICIs treatment and subsequent follow-up.

Exclusion Criteria:

* Individuals involved in the planning or implementation of the study;
* Concurrent use of other tumor treatment modalities during the study, including but not limited to: chemotherapy, radiotherapy, immunotherapy, microbial therapy, traditional Chinese medicine, and other investigational therapies;
* History of bilateral ovarian-related surgery;
* Patients with prior radiotherapy or chemotherapy causing irreversible damage to ovarian function;
* Individuals with known allergy to ICIs or their components;
* Patients with known non-response to immunomodulatory therapy;
* Patients with unexplained menstrual irregularities or long-term hormone medication use;
* Patients with chronic gastrointestinal disease or known dysbiosis (e.g., Crohn's disease, ulcerative colitis);
* Patients who frequently consume fermented foods;
* Patients who underwent major surgery within 3 weeks prior to study initiation or have not yet recovered from surgery;
* Subjects with other malignancies within the past 3 years;
* Patients with severe, uncontrolled medical conditions or those deemed by the investigator to be generally unsuitable for study participation, including but not limited to: active viral infections such as HIV, hepatitis B, hepatitis C; severe cardiovascular disease, uncontrolled ventricular arrhythmias, myocardial infarction within the past 3 months; uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or other psychiatric conditions affecting informed consent; uncontrolled hypertension despite medication; immunodeficiency (excluding splenectomy) or other conditions the investigator deems likely to expose the subject to high toxicity risk;
* Any history or current clinical evidence suggesting potential for confounding study results, compromising patient compliance throughout the study, or acting against the patient's best interests;
* Receipt of platelet or red blood cell transfusion within 3 days prior to initiation of study drug treatment;
* Pregnant or lactating patients, or patients planning pregnancy during the study period.
* Clinically unresolved prior treatment toxicity (≥ Grade 2, excluding alopecia, neuropathy, lymphopenia, or skin hypopigmentation);

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients with malignant tumors scheduled to receive ICI or combination therapy including ICI at the Department of Biological Therapy, West China Hospital, Sichuan University between September 2025 and May 2026
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Follicle-stimulating hormone | At the enrollment and the end of Cycle 6( each cycle is 28 days)
  Serum levels of Follicle-stimulating hormone
Luteinizing hormone | At the enrollment and the end of Cycle 6( each cycle is 28 days)
  Serum levels of Luteinizing hormone
Estradiol | At the enrollment and the end of Cycle 6( each cycle is 28 days)
  Serum levels of Estradiol
Progesterone | At the enrollment and the end of Cycle 6( each cycle is 28 days)
  Serum levels of Progesterone
Anti-Müllerian hormone | At the enrollment and the end of Cycle 6( each cycle is 28 days)
  Serum levels of Anti-Müllerian hormone
Gut microbiota composition | At the enrollment and the end of Cycle 6 (each cycle is 28 days)
  Analyzing gut microbiota composition using metagenomic data from patient feces

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Serum levels of FSH, LH, E2, P, and AMH hormones, along with fecal metagenomic sequencing data from patients, will be publicly shared at NCBI database.
Time Frame: IPD will be made available for sharing upon completion of the study.